CLINICAL TRIAL: NCT05182112
Title: Phase I Study of Precision CRT for Liver-Dominant Metastatic Pancreatic Cancer with Homologous Recombination Deficiency (PreCISeRT)
Brief Title: Radiation Therapy (RT) and Chemotherapy for the Treatment of Pancreatic Cancer with Homologous Recombination Deficiency That Has Spread to the Liver
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-443
Record Dates: First submitted 2021-12-20; First posted 2022-01-10 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Pancreatic Cancer
Keywords: Metastatic Pancreatic Cancer; Homologous Recombination Deficiency; Radiation Therapy (RT); 21-443
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Cisplatin

STUDY DESIGN:
Intervention Model Description: This is a phase I rolling 6 design dose escalation study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Radiation Therapy (RT) and Chemotherapy (Experimental): Upon enrollment in the study, patients will undergo radiation simulation. Protocol therapy will start upon completion of RT planning (1-2 weeks). Chemoradiation will be initiated 1-2 weeks later depending on RT planning and consist of whole liver irradiation (WLI).
  Interventions: Radiation: Whole liver irradiation (WLI); Drug: Gemcitabine and Cisplatin

INTERVENTIONS:
Radiation: Whole liver irradiation (WLI) — Whole liver irradiation (WLI) to a total dose 1800cGy in 10 fractions will be given over 2 weeks with simultaneously integrated boost (SIB) to deliver focal doses of 3600cGy (dose level 1) and 4800cGy (dose level 2) to select gross lesions. SIBl dose assignment will be according to the dose escalation scheme, with all patients in dose level 1 receiving boost of 3600cGy to select lesions and those in dose level 2 receiving boosts of 4800cGy to select lesions. At least one lesion will be selected for dose escalation.
Drug: Gemcitabine and Cisplatin — Patients will start cisplatin 10 mg/m2 and gemcitabine 600 mg/m2 intravenously q2 weeks for 1 cycle while undergoing simulation and radiation treatment planning procedures. After completion of CRT, adjuvant cisplatin 25 mg/m2 and gemcitabine 600 mg/m2 q2 weeks will be continued until progression or unacceptable toxicity.

SUMMARY:
The researchers are doing this study to test the combination of radiation therapy (RT) and low dose chemotherapy in people with metastatic pancreatic cancer that has a homologous recombination deficiency (HRD) and has spread to the liver. The researchers will try to find the highest safe and effective dose of individualized dose-painted RT that can be given to the liver when combined with standard low dose chemotherapy. The conformal dose painted RT treatment plan will include higher doses of radiation to the areas of the liver where tumors can be seen, and a lower dose to the entire liver. The study will also look at blood samples from participants to learn why some people may respond to study treatment (whole liver RT in combination with low dose chemotherapy) better than others.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the pancreas metastatic to the liver (liver metastases confirmed pathologically or radiographic liver lesions most consistent with metastases in a patient with pathologically proven pancreatic adenocarcinoma)
* Germline or biallelic somatic pathogenic mutations in the core HR genes including BRCA1, BRCA2, PALB2 and ATM genes are required for dose escalating cohort. Pathogenic germline or biallelic somatic alterations in other HR genes including (BAP1, BARD1, BLM, BRIP1, CHEK2, FAM175A, FANCA, FANCC, NBN, RAD50, RAD51, RAD51C, RTEL1) are allowed in the expansion cohort. Confirmation of the required mutations can be from MSK IMPACT or any other approved germline genetic testing for eligibility purposes.
* ≥1 liver lesion(s) measurable on a contrast-enhanced liver CT, MRI or PET/CT performed within 6 weeks prior to study entry. Any tumor location within the liver is allowed
* At least 1 liver metastasis measuring ≤ 7 cm
* Extrahepatic disease outside the liver is permitted if the hepatic disease is judged to be life-limiting (1-2 sites of disease are allowed, including lung and non-regional nodes, up to and including 5 individual lesions)
* Age ≥18
* ECOG 0-2
* Any prior chemotherapy therapy is allowed including prior treatment with platinum containing chemotherapy and irrespective of response to prior therapy
* Prior treatment with FDA-approved or investigational biologics or novel molecularly targeted therapies, including oral or IV formulations, are permitted. Patients must be off prior targeted therapy for at least 14 days or 4 half-lives prior to the initiation of the study treatment
* Use of an effective means of contraception in men and women of child-bearing potential
* Adequate organ and marrow function within 14 days prior to study entry, defined as:
* Absolute neutrophil count (ANC)>1000/mm3
* Hemoglobin >9 gm/dl (Note: The use of transfusion or other intervention to achieve Hgb > 9.0 g/dl is acceptable.)
* Platelets >100,000/mm3
* Serum creatinine <1.5 mg/dl OR creatinine clearance of >50 cc/min
* Total bilirubin < 1.8 mg/dL
* Prothrombin time/INR < 1.7
* Albumin ≥ 28 g/L
* AST and ALT < 3 times ULN
* ALP < 2.5 times ULN

Exclusion Criteria:

* Prior invasive malignancy, except non-melanoma skin cancer, unless disease free for a minimum of 3 years
* Prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields.
* History of underlying liver disease, including but not limited to cirrhosis, hepatitis or hemochromatosis
* History of major liver resection
* Variants of unknown significance (VUS) in core or non-core HR genes will be excluded
* Severe, active co-morbidity, defined as follows:

  * Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months
  * Transmural myocardial infarction within the last 6 months
  * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration
  * Chronic Obstructive Pulmonary Disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration
* Clinical ascites.
* Single right kidney. (A single left kidney is allowed)
* Absolute contraindication to cisplatin including severe hypersensitivity
* Pregnancy, nursing women, or women of childbearing potential, and men who are sexually active and not willing/able to use medically acceptable forms of contraception; this exclusion is necessary because the treatment involved in this study may be significantly teratogenic.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2021-12-20 (Actual); Primary Completion 2024-11-04 (Actual); Study Completion 2024-11-04 (Actual)

PRIMARY OUTCOMES:
determine the maximum tolerated dose of focal simultaneously integrated boost (SIB) | 1 year
  we will use a rolling 6 dose-escalation design which allows for accrual of two to six patients concurrently onto a dose level (hence tends to shorten the study conduct timeline) based on the number of patients currently enrolled and evaluable, the number experiencing dose-limiting toxicity (DLT), and the number still at risk of developing a DLT.

CONTACTS AND LOCATIONS:
Overall Officials: Marsha Reyngold, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (All Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (All Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (All Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk - Commack (All Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (All Protocol Activities), East White Plains, New York
  - Memorial Sloan Kettering Cancer Center (All protocol activities), New York, New York
  - Memorial Sloan Kettering Nassau (All Protocol Activities), Rockville Centre, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm